CLINICAL TRIAL: NCT06261112
Title: The Effect of the Use of Kaleidoscope on Pain and Fear in the Plastering Process of Fracture Emergencies
Brief Title: The Effect of Using a Kaleidoscope on Fear and Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mihriban Culha (Other)
Responsible Party: Sponsor-Investigator, Mihriban Culha, study director, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.01.11/285
Record Dates: First submitted 2024-01-04; First posted 2024-02-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Fracture; Complication Orthopedic Procedure
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Parallel Assigment
Who Masked: Investigator
Masking Description: single /investigatör)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group kaleideskope, pain and fear
  Interventions: Other: kaleidescope
- No intervention group (No Intervention): No intervention group Control not pain and fear

INTERVENTIONS:
Other: kaleidescope — used to kaleideskope
  Arms: Experimental group

SUMMARY:
The research was conducted in randomized controlled experimental type between May 2022 and December2023. The universe of the research consisted of children and their parents who were diagnosed with a fracture, applied to the Orthopedic outpatient clinic and Emergency department of the Erzurum Ataturk University Health Research and Application Center and referred to the Orthopedic clinic, and decided to undergo a cast procedure for treatment. The sample of the research consisted of a total of 70 children and their parents, including 35 control groups and 35 kaleidoscope groups, who met the research criteria from this universe. The children in the kaleidoscope group were shown the kaleidoscope. No intervention other than routine application was applied to the control group. "Introductory Information Form", "Wong-Baker Facial Expressions Rating Scale and Child Fear Scale were used in the collection of data.

DETAILED DESCRIPTION:
Type of Study: The study was designed as a randomized controlled experimental study. Place and Time of Research:

The research was conducted between March 2022 and December 2023 as a randomized controlled experimental study. The study population consisted of patients who sought treatment at the Orthopedics Polyclinic and Emergency Department of Erzurum Atatürk University Health Research and Application Center. These patients were referred to the orthopedics clinic and diagnosed with fractures, such as humerus, wrist, finger, tibia, femur, and ankle fractures, for which plastering was performed as treatment. Specifically, the study included children aged 6 to 12 years. The sample size for the study was determined through a power analysis and ultimately consisted of a total of 70 children, with 35 children assigned to both the control group and the kaleidoscope group. The children in the kaleidoscope group were exposed to a kaleidoscope, while the control group received no intervention beyond routine medical practice. To collect data, the researchers utilized an "Introductory Information Form," the "Wong-Baker Faces Pain Rating Scale," and the "Children Fear Scale." The data were analyzed using percentage distributions, mean, standard deviation, chi-square test, and independent groups t-test. Throughout the research, ethical principles were strictly followed.

ELIGIBILITY:
Inclusion Criteria:

* Being a child in the 6-12 age group,
* The child's willingness to participate in the study,
* The parent's volunteering to participate in the study,
* Absence of intellectual disability of the child and parent,
* The child and the parent speak Turkish and are open to communication.

Exclusion Criteria:

* The child has a chronic disease that can cause pain,
* The child has used analgesics within 24 hours before admission to the hospital,
* The child has visual impairment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Child Fear Scale (CFS) | 12 MONTHS
  The Child Fear Scale was developed by McMurty et al. in 2011 to measure fear in children undergoing painful medical procedures. The Child Fear Scale is a 0-4 Likert type scale showing five different faces, ranging from neutral (0=n0 concern et all) to fearful (4=severe anxietly).

SECONDARY OUTCOMES:
Facial Expressions Rating Scale | 12 MONTHS
  This visual facial scale is a practical method to assess rhe level of anxiety within a situation. There are six facial expressions, ranging from very happy to very unhappy and children are asked to choose the one that comes closest to how they feel at that moment. The most positive face is scored as "0" and the most negative face as scored as "5".

CONTACTS AND LOCATIONS:
Overall Officials: Mihriban ÇULHA, Principal Investigator — Mihriban ÇULHA, graduate student ,Ataturk University; Mihriban ÇULHA, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE ARTİCLE IS INTENDED TO BE SHARED AFTER PUBLİCATİON